CLINICAL TRIAL: NCT03834623
Title: A Phase II Biomarker Trial of Avadomide (CC-122) in Combination With Nivolumab in Advanced Melanoma
Brief Title: Avadomide (CC-122) in Combination With Nivolumab in Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19706
Record Dates: First submitted 2019-02-04; First posted 2019-02-08 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: melanoma; skin
MeSH Terms: conditions — Melanoma | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-122 Plus Nivolumab (Experimental): Participants will take CC-122 orally at 2mg daily for 5 consecutive days every 7 days, with intravenous nivolumab (240mg) in days 1 and 15 within a 28-day cycle.
  Interventions: Drug: CC-122; Drug: Nivolumab

INTERVENTIONS:
Drug: CC-122 — Oral CC-122 at 2 mg daily, 5 days out of 7
  Other Names: Avadomide
Drug: Nivolumab — 240 mg Nivolumab intravenously days 1 and 15 in each 28 day cycle
  Other Names: Opdivo

SUMMARY:
This study is to find out if the combination of CC-122 (an investigational agent) and Nivolumab will enhance the anti-cancer activity and prevent T-cell exhaustion (T-cells are responsible for maintaining the body's immune response).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic melanoma of cutaneous, mucosal, conjunctival, or unknown origin. Uveal melanoma is not permitted. Cohort 1: Naïve to anti-PD1 therapy Cohort 2: Progressed on previous anti-PD1 therapy. Subjects who have received anti-PD1 therapy in the adjuvant setting for previously resected melanoma are eligible for this cohort provided they have not received any intervening systemic therapy for the relapse
* Be willing and able to provide written informed consent for the trial.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Females of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Females of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study 28 days after last dose of avadomide or 5 months after the last dose of nivolumab, whichever is longer. Females of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.
* Males should agree to use an adequate method of contraception starting with the first dose of study therapy through 3 months after the last dose of avadomide or 7 months after last dose of nivolumab, whichever is longer.
* Adequate organ function

Exclusion Criteria:

* Has received an investigational drug or other anti-cancer therapy within 3 weeks of the first dose of treatment or < 5 half-lives of that agent, whichever is shorter. Any toxicity from prior therapy must have recovered to < grade 1.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (only exception to this is the need for steroids for CNS metastases; see #6 below). Inhaled, intra-articular, or topical steroids are permissible.
* Has a history of hypersensitivity to nivolumab.
* Has a known additional malignancy that is progressing or requires active treatment, the lack of which would pose a risk to the health of the subject, in the opinion of the investigator.
* Has known symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable without evidence of progression by imaging for at least four weeks after definitive intervention and using no more than the equivalent of dexamethasone 2mg/d for the management of vasogenic edema, if necessary. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy [</= 10 mg/d equivalent of prednisone] for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with previous grade III/IV toxicity from immunotherapy that led to treatment discontinuation are excluded.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the investigator.
* Is pregnant or breastfeeding.
* Has a known history of Human Immunodeficiency Virus (HIV), active Hepatitis B or Hepatitis C.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Khushalani, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Anti-PD1 Naive: Anti-PD1 naive participants will take CC-122 orally at 2mg daily for 5 consecutive days every 7 days, with intravenous nivolumab (240mg) in days 1 and 15 within a 28-day cycle.
  CC-122: Oral CC-122 at 2 mg daily, 5 days out of 7 Nivolumab: 240 mg Nivolumab intravenously days 1 and 15 in each 28 day cycle
- Cohort 2: Anti-PD1 Refractory: Anti-PD1 refractory participants will take CC-122 orally at 2mg daily for 5 consecutive days every 7 days, with intravenous nivolumab (240mg) in days 1 and 15 within a 28-day cycle.
  CC-122: Oral CC-122 at 2 mg daily, 5 days out of 7 Nivolumab: 240 mg Nivolumab intravenously days 1 and 15 in each 28 day cycle
Period: Overall Study
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Started | 11 | 12
Completed | 11 | 11
Not Completed | 0 | 1
Not completed — Progression | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 7 | 8 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate of CC-122 in Combination With Nivolumab
Description: Objective Response Rate of CC-122 in combination with Nivolumab in both anti-PD1 therapy naive advanced melanoma as well as anti-PD1 therapy refractory melanoma (primary refractory or progressing after an initial response or stable disease)
Time Frame: Up to 52 weeks
Measure: Median (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 11 | 12
proportion of participants | .545 [.23 to .83] | 0 [0 to 0]

2. Secondary Outcome: Number of Participants Who Experience Treatment Related Adverse Events
Description: All Adverse Events and Serious Adverse events will be collected and collated according to grade and frequency. This will include all events considered possibly, probably or definitely related to study therapy.
Time Frame: Up to 52 weeks
Measure: Number; unit: participants
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 11 | 12
participants | 11 | 12

3. Secondary Outcome: Tumor Response
Description: Tumor response will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and and iRECIST (Response Evaluation Criteria in Solid Tumors in immunotherapy) guidelines v1.1. Results will be indicated as number of participants with evaluable tumor response.
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 11 | 12
Participants | 11 | 12

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival will be calculated from the start of study therapy till the first documentation of disease progression, death, or change of treatment. Subjects receiving ongoing therapy at the time of data analysis will be censored
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 11 | 12
months | NA [5.7 to NA] — Not reached, participants not followed for survival beyond 24 months. | 2.7 [2.7 to NA] — Not reached, participants not followed for survival beyond 24 months.

5. Secondary Outcome: Overall Survival
Description: Overall survival will be calculated from the start of therapy till death from any cause. Subjects alive at the time of data analysis will be censored.
Time Frame: Up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
Number analyzed (Participants) | 11 | 12
months | NA [24.0 to NA] — Not reached, participants not followed beyond 24 months | 11.5 [5.5 to NA] — Not reached, participants not followed beyond 24 months

ADVERSE EVENTS:
Time Frame: Adverse events collected from time of informed consent to 30 days after study participation, approximately 2.5 years.
Arm/Group | Cohort 1: Anti-PD1 Naive | Cohort 2: Anti-PD1 Refractory
All-Cause Mortality (participants affected / at risk) | 0/11 | 3/12
Serious Adverse Events (participants affected / at risk) | 3/11 | 6/12
Other Adverse Events (participants affected / at risk) | 11/11 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Anti-PD1 Naive (N=11) | Cohort 2: Anti-PD1 Refractory (N=12)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) — Pnemonia
Cardiac troponin T increased (Investigations) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — coronary artery bypass graft surgery
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 0 (0) | 1 (1) — Diverticulitis
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Anti-PD1 Naive (N=11) | Cohort 2: Anti-PD1 Refractory (N=12)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (3) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (9) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (4) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (16) | 10 (16)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 5 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 5 (18) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (3) | 0 (0)
Cardiac troponin T increased (Investigations) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Chills (General disorders) | 1 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Creatinine increased (Investigations) | 2 (9) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (6) | 4 (11)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Dizziness (Nervous system disorders) | 5 (7) | 4 (4)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 4 (9)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 3 (5)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Endocrine disorders - Other (Endocrine disorders) | 1 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eye disorders - Other (Eye disorders) | 2 (11) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (18) | 8 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 1 (3)
Flushing (Vascular disorders) | 3 (3) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (3) | 3 (5)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 5 (6) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 2 (2) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (13) | 5 (10)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (11) | 6 (11)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (8) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (9) | 5 (6)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 6 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Investigations - Other (Investigations) | 10 (51) | 9 (22)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Lethargy (Nervous system disorders) | 1 (1) | 2 (2)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 2 (3)
Lung infection (Infections and infestations) | 1 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (16) | 6 (7)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (5)
Neck edema (General disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 4 (5)
Nervous system disorders - Other (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (42) | 4 (8)
Non-cardiac chest pain (General disorders) | 2 (3) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (8) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (2) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 2 (11) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (17) | 7 (8)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 3 (4)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 (15) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 2 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testosterone deficiency (Endocrine disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (3)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (4)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (2)
Vascular disorders - Other (Vascular disorders) | 1 (2) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)
Weight gain (Investigations) | 1 (2) | 2 (3)
Weight loss (Investigations) | 3 (4) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 7 (33) | 5 (8)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03834623/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03834623/ICF_002.pdf